CLINICAL TRIAL: NCT02859038
Title: Study of Upfront Surgery Versus Neoadjuvant Chemotherapy Followed by Interval Debulking Surgery for Patients With Stage IIIC and IV Ovarian Cancer
Brief Title: Study of Upfront Surgery Versus Neoadjuvant Chemotherapy in Patients With Advanced Ovarian Cancer (SUNNY)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGOG OV4B; SOC-2 (Other: Shanghai Gynecologic Oncology Group)
Record Dates: First submitted 2016-07-23; First posted 2016-08-08 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Upfront cytoreductive surgery (Experimental): Upfront cytoreductive surgery with a maximal cytoreduction of complete gross resection within 3 weeks after biopsy, followed by at least 6 cycles of adjuvant chemotherapy.
  Interventions: Procedure: Upfront cytoreductive surgery
- Neoadjuvant chemotherapy (Active Comparator): neoadjuvant chemotherapy with 3 cycles of chemotherapy, then followed by interval debulking surgery. The maximal time interval between course 3 chemotherapy and IDS is 6 weeks. And then 3 cycles of adjuvant chemotherapy.
  Interventions: Procedure: Interval debulking surgery

INTERVENTIONS:
Procedure: Upfront cytoreductive surgery — Upfront cytoreductive surgery with a maximum cytoreduction, then followed by 6 cycles of Paclitaxel 175mg/m2 or Docetaxel 60-75 mg/m2 plus Carboplatin AUC (area under the curve) 5
  Other Names: Primary debulking surgery, PDS
  Arms: Upfront cytoreductive surgery
Procedure: Interval debulking surgery — 3 cycles of Paclitaxel 175mg/m2 or Docetaxel 60-75 mg/m2 plus Carboplatin AUC (area under the curve) 5, Interval debulking surgery with a maximal cytoreduction of complete gross resection, then followed by another 3 cycles of chemotherapy
  Other Names: NACT-IDS
  Arms: Neoadjuvant chemotherapy

SUMMARY:
The purpose of this study is to answer the fundamental question, should the physicians choose Surgery or Chemotherapy (SOC-2) in advanced ovarian cancer?

DETAILED DESCRIPTION:
OBJECTIVES: Compare the efficacy and safety in patients with AJCC TNM stage IIIC or IV epithelial ovarian cancer, fallopian tube cancer, or peritoneal carcinoma treated with neoadjuvant chemotherapy followed by interval debulking surgery versus upfront surgery.

OUTLINE: This is a randomized phase III multicenter study. Patients will receive upfront maximal cytoreductive surgery followed by at least 6 cycles of adjuvant chemotherapy or 3 cycles of neoadjuvant chemotherapy followed by interval debulking surgery, and then at least 3 cycles of adjuvant chemotherapy.

Patients are followed every 3 months within the first 5 years, and then every 6 months.

PROJECTED ACCRUAL: A total of 488 patients will be accrued for this study within 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥ 18 years.
2. Pathologic confirmed stage IIIC and IV epithelial ovarian cancer, fallopian tube cancer or primary peritoneal carcinoma (diagnosis by biopsy or fine needle aspiration*). Laparoscopic biopsy with pictures is recommended.

   * If fine needle aspiration showing an adenocarcinoma, patients should satisfy the following conditions: a. the patient has a pelvic mass, and b. omental cake or other metastasis larger than 2 cm in the upper abdomen, or pathologic confirmed extra-abdominal metastasis, and c. serum CA125/CEA ratio>25. If serum CA125/CEA ratio<25 or malignancies of other origins, such as breasts and digestive tract, are suspected from symptoms, physical examinations or imaging diagnosis, endoscopy or ultrasonography should be done to exclusive metastasis ovarian cancer.
3. ECOG performance status of 0 to 2.
4. ASA score of 1 to 2.
5. Adequate bone marrow, liver and renal function to receive chemotherapy and subsequently to undergo surgery:

   1. white blood cells >3,000/µL, absolute neutrophil count ≥1,500/µL, platelets ≥100,000/µL, hemoglobin ≥9 g/dL,
   2. serum creatinine <1.25 x upper normal limit (UNL) or creatinine clearance ≥60 mL/min according to Cockroft-Gault formula or to local lab measurement,
   3. serum bilirubin <1.25 x UNL, AST(SGOT) and ALT(SGPT) <2.5 x UNL.
6. Comply with the study protocol and follow-up.
7. Written informed consent.

Exclusion Criteria:

1. Patients with non-epithelial tumors as well as borderline tumors.
2. Mucinous ovarian cancer.
3. Low grade ovarian cancer.
4. Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ.
5. Any other concurrent medical conditions contraindicating surgery or chemotherapy that could compromise the adherence to the protocol.
6. Other conditions, such as religious, psychological and other factors, that could interfere with provision of informed consent, compliance to study procedures, or follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2016-08; Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Participants will be followed for at least 5 years after randomization or until death
  The time from entry into the study to any cause of death.

SECONDARY OUTCOMES:
Progression-free survival | Participants will be followed for at least 5 years after randomization or until death
  The time from entry into the study to the diagnosis of the first progression or recurrence or death, whichever occurs first.
Post-operative complications | Participants will be followed up to 6 months after randomization
  The surgical complications will be evaluated at 30-day after upfront cytoreductive surgery or interval debulking surgery.
Quality of life assessments | Participants will be followed for at least 5 years after randomization or until death
  QOQ-C30,FACT-O( baseline; 6months, 12 months and 5 years after randomization)
Accumulated treatment-free survival (TFSa) | Participants will be followed for at least 5 years after randomization or until death
  The overall survival time minus the total treatment time of surgery and chemotherapy after randomization, but maintenance of targeted agents is considered off-treatment.
Time to first subsequent anticancer therapy (TFST) | Participants will be followed for at least 5 years after randomization or until death
  The date of randomization until the starting date of the first subsequent anticancer therapy or death, whichever occurs first. Maintenance treatments following a cytostatic treatment are NOT considered separate treatment lines.
Time to second subsequent anticancer therapy (TSST) | Participants will be followed for at least 5 years after randomization or until death
  The date of randomization until the starting date of the second subsequent anticancer therapy or death, whichever occurs first. Maintenance treatments following a cytostatic treatment are NOT considered separate treatment lines.
The pattern of the first relapse | Participants will be followed for at least 5 years after randomization or until death
  The number and sites of the first relapse, including pelvic, abdominal, retroperitoneal lymph nodes, distant metastases and ascites will be compared between the two groups.
The rate of 5-year progression-free survival | Participants will be followed for at least 5 years after randomization or until death
  The rate of the patients without progression or recurrence or death at 5 years.
Outcomes of pulmonary embolism | Participants will be followed for at least 5 years after randomization or until death
  The incidence of pulmonary embolism prior to primary treatment in the ITT and hospital populations. Its effect on survival between groups in the ITT and hospital populations.

CONTACTS AND LOCATIONS:
Overall Officials: Rongyu Zang, MD,PHD, Principal Investigator — Fudan University Shanghai Zhongshan Hospital
Locations (8):
- China (6):
  - Sun Yet-Sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Hunan Provincial Hospital, Changsha
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiang R, Zhu J, Kim JW, Liu J, Kato K, Kim HS, Zhang Y, Zhang P, Zhu T, Aoki D, Yu A, Chen X, Wang X, Zhu D, Zhang W, Jia H, Shi T, Gao W, Yin S, Feng Y, Xiang L, Okamoto A, Zang R. Study of upfront surgery versus neoadjuvant chemotherapy followed by interval debulking surgery for patients with stage IIIC and IV ovarian cancer, SGOG SUNNY (SOC-2) trial concept. J Gynecol Oncol. 2020 Sep;31(5):e86. doi: 10.3802/jgo.2020.31.e86. PMID 32808504
- See also: Shanghai Gynecologic Oncology Group — http://www.ShanghaiGOG.org